CLINICAL TRIAL: NCT00318903
Title: A Phase II Study of Irinotecan and Taxotere With Concurrent Radiotherapy as a Preoperative Treatment in Resectable Esophageal Cancer
Brief Title: Irinotecan and Taxotere With Radiotherapy as Preoperative Treatment in Resectable Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Pharmacia and Upjohn (Industry)
Responsible Party: Principal Investigator, Michael James Bertram, Proffessor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F001130016; UAB 0032 (Other: institutional study protocol number)
Record Dates: First submitted 2006-04-13; First posted 2006-04-27 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Esophageal Cancer; Cancer of the Esophagus; Esophagus Cancer; Esophageal Neoplasm; Cancer of Esophagus
Keywords: Chemotherapy for cancer of the esophagus; Radiotherapy for cancer of the esophagus; Surgery for cancer of the esophagus; Chemotherapy, radiotherapy, surgery for esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Irinotecan; Pharmaceutical Preparations; Docetaxel; Radiotherapy; Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Taxotere/Irinotecan (Experimental): Taxotere and Irinotecan is given intravenously for 3 consecutive weeks with a one-week break before radiotherapy for 5-6 weeks. A combination of Taxotere and Irinotecan will then be administered simultaneously with the radiotherapy.
  Interventions: Drug: Irinotecan (drug); Drug: Taxotere (drug); Procedure: Radiotherapy (procedure); Procedure: Esophagectomy (procedure)

INTERVENTIONS:
Drug: Irinotecan (drug) — 50 mg/m2 of Irinotecan will be administered intravenously over 60-90 minutes following a Taxotere infusion each week for 3 weeks. After a break, Irinotecan will then be given for 3 consecutive weeks at 45 mg/m2 in conjunction with radiotherapy.
  Other Names: Camptosar
Drug: Taxotere (drug) — Taxotere at 35 mg/m2 is given intravenously over 1 hour each week for three consecutive weeks. After a one-week break, patients will receive Taxotere at a 25 mg/m2 dose for the first three weeks of a 5-6 week radiotherapy regimen.
  Other Names: Docetaxel
Procedure: Radiotherapy (procedure) — Radiotherapy will be given in 28 fractions over 5-6 weeks at 1.8 Gy per fraction for a total of 50.4 Gy. This will begin concurrently with chemotherapy on Day 29 of treatment.
Procedure: Esophagectomy (procedure) — After approximately 14 weeks of treatment, the patient will be evaluated for surgery. Only those who have achieved a good response will be eligible.

SUMMARY:
There is a need for more effective therapy for patients following surgery for esophageal carcinoma. Docetaxel and Irinotecan, independent of each other, have demonstrated activity in this disease. There is interest in the combination of these two active agents plus radiotherapy.

DETAILED DESCRIPTION:
The high rate of local and distant failure following surgery for esophageal carcinoma necessitates a more effective therapy for these patients. The merit of neoadjuvant chemotherapy is early management of micrometastatic disease and radiosensitization. A longstanding regimen, 5-FU and Cisplatin, have failed to produce a substantial survival benefit, but the approach has resulted in pathologic complete responses prior to surgical eradication of the diseased organ. This raises questions of organ preservation in some patients. Docetaxel and Irinotecan have both demonstrated independent activity in this disease and are radiosensitizers. In this study, Docetaxel and Irinotecan will be given together weekly for 3 consecutive weeks in an attempt to decrease the recurrence of systemic disease, and this will be followed by giving each agent independently with radiation therapy to decrease the local relapse rate and independently measure the toxicity of each with radiation. Following completion of chemoradiotherapy, the patients will undergo resection and be evaluated for the pathologic response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of adenocarcinoma/squamous cell carcinoma of the esophagus. Patients should be considered resection candidates, Clinical Stages II- IV (For GE junction tumors 50% of the tumor must be within the esophagus)
* Age 19 years
* Male or female gender (not pregnant or lactating). If the subject is fertile, use of medically acceptable contraception will be required, and women with reproductive potential shall have a negative pregnancy test.
* Patient should be able to understand and offer signed written informed consent prior to study entry.
* No prior receipt of surgery, chemotherapy, radiotherapy or immunotherapy.
* Patients must demonstrate a ECOG P.S. ≤ 1
* Minimum life expectancy of 12 weeks
* End Organ function must be adequate meeting the below criteria at baseline:

WBC 3000/mm3, ANC 1500/mm3 , Hgb 9.0 g/dL, PLT 100,000mm3 Normal serum creatinine ( 1.5 mg/dL) Total Bilirubin ULN, Transaminases (SGOT and/or SGPT) may be up to 1.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is < ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are < ULN.

PT/PTT below the upper limit of normal (patients may be on 1mg of Coumadin for line patency) Peripheral neuropathy must be < Grade 1

Exclusion Criteria:

* Diagnosis of active, invasive (treated in past 5 years) concomitant malignancy except non-melanotic skin cancer
* Patients must be fully recovered from any reversible side effects of prior intervention
* Presence of an underlying disease state associated with impairment of performance status
* New York Heart Association Class IV congestive heart failure
* Limited mental capacity or language skills to the extent simple instructions cannot be followed or information regarding adverse events cannot be provided

History of non-compliance with prescribed medical care.

* Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80 must be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-01; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The determination of pathologic response in patients who undergo surgical resection. | Approximately 14 weeks before eligible patients have surgery

SECONDARY OUTCOMES:
To assess the overall survival, time to treatment failure, and quality of life in patients who receive any therapy | Approximately 4 months
To assess the toxicities associated with this treatment and any impact on surgery. | Approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: James A. Posey, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States